CLINICAL TRIAL: NCT00942214
Title: Biomarkers Associated With Response to Natalizumab in Multiple Sclerosis Patients. A Prospective Multicentric Open Label Phase IV Study
Brief Title: Biomarkers and Response to Natalizumab for Multiple Sclerosis Treatment
Acronym: Bionat2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: LESTIME Elodie, University Hospital, Toulouse
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0811001
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; natalizumab; pharmacogenomics
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Natalizumab — 300mg, IV, every 4 weeks
  Other Names: Tysabry (brand name)

SUMMARY:
Information from blood samples may help us for choosing the best treatment in future personalized medicine. Natalizumab (NTZ) a current treatment for MS can be used as a second line therapy if a suboptimal response to disease modifying drugs. When to introduce NTZ is not consensual. The investigators hypothesized that biological information could rationalize choice and thus designed a prospective open label trial to test biological markers before treatment.

DETAILED DESCRIPTION:
Current state of knowledge of the topic of the project and The general interest of the project; Pharmacogenomic aims to determine biomarkers related to treatment response, a step toward patient-tailored medicine. Natalizumab, a monoclonal antibody has just received the EMEA approval for MS patients who do not respond to interferon treatment or who experience a severe disease course. Efficacy of the drug is outstanding with 37% of the patients completing the "disease free" definition after 2 years (7% in placebo group). On the other hand, natalizumab may be associated with severe adverse events such as progressive multifocal leucoencephalopathy and high costs. Overall, this emphasizes the need beyond current approval criteria to identify those patients with the best efficacy to safety ratio, a major public health issue.

Scientific aims The primary scientific aim is to define biomarkers that would allow predicting long term response to natalizumab.

Methodology; The investigators plan to conduct a 5 years study to search for the best predicting factors at the beginning of treatment and after 2 years. In this grant application the investigators will perform a multivariate analysis of clinical, MRI, and biological markers (neutralizing antibody, DNA, and mRNA expression) from baseline to 2 years. For feasibility reasons, long term follow up (5 years) and proteomics study will be performed in a second stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 55 years.
* Diagnosis of relapsing multiple sclerosis according to McDonald criteria.
* EDSS score of 0 to 5.0 on the EDSS scale. One of the following 2 items:

  1. Patients who have failed to respond to a full and adequate course of a beta-interferon. Patients have had at least 1 relapse in the previous year while on therapy, and have at least 9 T2-hyperintense lesions in cranial MRI or at least 1 Gadolinium-enhancing lesion.
  2. Patients with rapidly evolving severe relapsing remitting multiple sclerosis, defined by 2 or more disabling relapses in one year, and with 1 or more Gadolinium enhancing lesions on brain MRI or a significant increase in T2 lesion load as compared to a previous recent MRI.

Exclusion Criteria:

* Hypersensitivity to natalizumab or to any of the excipients.
* Progressive Multifocal Leukoencephalopathy (PML).
* Increased risk of opportunistic infections, including immunocompromised patients (including those currently receiving immunosuppressive therapies or those immunocompromised by prior therapies, e.g. mitoxantrone or cyclophosphamide within 1 year before Tysabri.
* Combination with beta-interferons or glatiramer acetate.
* Known active malignancies, except for patients with cutaneous basal cell carcinoma.
* Children and adolescents.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
haplotypic frequency difference between responders and non-responders | 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David Brassat, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- service de neurologie, hôpital Purpan, Toulouse, France